CLINICAL TRIAL: NCT04526600
Title: Can Fidgeting Lead to Enhanced Attention and Emotional Regulation in ADHD?
Brief Title: Fidgeting and Attentional and Emotional Regulation in ADHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1607722
Record Dates: First submitted 2020-08-11; First posted 2020-08-26 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No fidget (No Intervention)
- With fidget (Experimental): The participant is given a specially designed fidget ball
  Interventions: Other: Fidget ball

INTERVENTIONS:
Other: Fidget ball — Access to a prototype 'smart' fidget ball with pressure sensors embedded, that produces touch traces and transmits real time data
  Arms: With fidget

SUMMARY:
This project will study how fidgeting relates to cognitive and emotional functioning in adults with attention-deficit/hyperactivity disorder (ADHD). It will determine, in a laboratory setting, whether movement and access to a "fidget device" providing sensory and motor stimulation can improve cognitive and emotional regulation (including on physiological measures) in adult ADHD. The investigators will also acquire pilot data for machine learning analyses to be used in future, large scale studies to identify gestures and touch characteristics associated with improved cognitive and emotional regulation to see if the data can predict and subsequently develop recommendations to improve performance and emotional control in natural settings (e.g., home, office, college classroom) for adult ADHD.

DETAILED DESCRIPTION:
Fidgeting is a highly common behavior, with excessive fidgeting associated with attention-deficit/hyperactivity disorder (ADHD). Studies from the investigator's laboratory and colleagues suggest physical movement can enhance cognitive performance in children with ADHD. Hyper-sensorimotor behavior may be related to impaired regulation of arousal in the noradrenergic and dopaminergic systems. This project will assess if frequency and characteristics of sensorimotor behavior relates to cognitive and emotional response in adults with ADHD, in a fine-grained manner, unlike other studies. The investigators will test if intrinsic fidgeting (Aim 1) and access to a specially designed fidget device (Aim 2) modulates behavioral and physiological response in cognitively and emotionally-demanding contexts. The hype of the commercially available fidget devices, its competitors and fidget spinners suggest it might, but there is no systematic evidence to inform consumers, a gap, the investigators aim to fill.

ELIGIBILITY:
Inclusion Criteria:

* ADHD
* History of fidgeting

Exclusion Criteria:

* Currently taking psychoactive medication, with the exception of stimulant medication for ADHD or medication that can affect heart rate;
* Presence of significant depression or psychotic disorders, autism, visual or hearing impairment or any other disorder that may interfere with task performance; and IQ below 85

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 109 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Processing speed | Day 1
  Paced Auditory Serial Addition Task (PASAT)
Working memory | Day 1
  List Sorting Test
Response inhibition | Day 1
  Flanker type test

SECONDARY OUTCOMES:
Physiological response as an index of emotional regulation | Approximately 45 minutes
  Heart rate variability and pre ejection period

CONTACTS AND LOCATIONS:
Overall Officials: Julie Schweitzer, Ph.D., Principal Investigator — UC Davis MIND Institute
Locations (1):
- UC Davis MIND Institute, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared via NDAR
Supporting Information: Study Protocol
Time Frame: Undecided, likely after publication date
Access Criteria: Will be through NDAR

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/can-fidgeting-lead-to-enhanced-attention-and-emotional-regulation-in-adhd-449990/